CLINICAL TRIAL: NCT05106101
Title: A Pilot/Phase 1, Interventional, Open-label, Multi-center Study to Assess the Safety and Efficacy of L-glutamine Treatment in Patients With Diverticulosis
Brief Title: L-glutamine Treatment in Patients With Diverticulosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emmaus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-DsD-002
Record Dates: First submitted 2021-09-22; First posted 2021-11-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-11

CONDITIONS: Diverticulosis, Colonic
MeSH Terms: conditions — Diverticulosis, Colonic | interventions — Glutamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-glutamine (Experimental): Participants received L-glutamine oral powder 15 grams twice daily for 48 weeks
  Interventions: Drug: L-glutamine

INTERVENTIONS:
Drug: L-glutamine — L-glutamine oral powder in 5 gram packet
  Other Names: oral L-glutamine

SUMMARY:
The purpose of the study is evaluate the safety and efficacy of L-glutamine as a treatment for patients with diverticulosis.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 4 weeks screening period to determine eligibility for study entry. At Week 0, patients who meet eligibility requirements will be given L-glutamine (15 grams, twice daily)

ELIGIBILITY:
Inclusion Criteria:

1. ≥50 years of age.
2. Uncomplicated diverticulosis confirmed by colonoscopy.
3. Colonoscopy indicates ≥5 colonic diverticula (pouches) in the descending/sigmoid colon and < approximately10 colonic diverticula (pouches) per segment (e.g. proximal descending, distal descending, proximal sigmoid, and distal sigmoid.)
4. If the patient is a female of child-bearing potential, she agrees to avoid pregnancy during the study and is willing and agrees to practice a recognized form of birth control during the course of the study (e.g., barrier, birth control pills, or abstinence).
5. Patients who have given their free and written informed consent.

Exclusion Criteria:

1. Acute diverticulitis (both complicated and uncomplicated).
2. Acute colitis
3. History of inflammatory bowel disease, colon resection, polyposis syndrome, severe strictures, and perforation.
4. Active bleeding
5. More than 40 diverticula
6. Chronic renal insufficiency
7. Chronic liver disease.
8. Patient is pregnant or lactating or has the intention of becoming pregnant during the study (if female of childbearing potential).
9. Inability to give a valid informed consent or to properly follow the protocol.
10. Patients with an active malignancy of any type, or a recent history of malignancy within the last 5 years.
11. Treated with an investigational medication/treatment within 30 days prior to the screening visit.
12. Currently enrolled in an Investigational study
13. Patient is currently taking or has been treated with any form of glutamine supplement within 30 days of the screening visit.
14. Previous difficulty pulling or passing of scope or difficulty completing colonoscopy.
15. There are factors that would, in the judgment of the investigator, make it difficult for the patient to comply with the requirements of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of colonic diverticula via colonoscopy at 6 and 12 months in patients with diverticulosis. | Baseline, 6 months and 12 months
  Number of diverticula for both the descending colon and sigmoid will be counted at baseline, at 6 months and at 12 months

SECONDARY OUTCOMES:
Change from baseline the size of colonic diverticula via colonoscopy at 6 and 12 months in patients with diverticulosis | Baseline, 6 month and 12 months
  Size of diverticula at the descending and sigmoid colon will be estimated as small only, large only, or both small and large, where large is defined as greater than 7 mm in diameter
Effect of oral L-glutamine on Hematological Parameters - Hemoglobin | Baseline to 48 weeks (12 months)
  Patient's hemoglobin will be collected at each visit
Effect of oral L-glutamine on Hematological Parameters - Hematocrit | Baseline to 48 weeks (12 months)
  Patient's hematocrit will be collected at each visit
Effect of oral L-glutamine on Vital Signs - Blood Pressure | Baseline to 48 weeks (12 months)
  Patient's blood pressure will be collected at each visit
Effect of oral L-glutamine on Vital Signs - Pulse Rate | Baseline to 48 weeks (12 months)
  Patient's pulse rate will be collected at each visit
Effect of oral L-glutamine on Vital Signs - Temperature | Baseline to 48 weeks (12 months)
  Patient's temperature will be collected at each visit
Effect of oral L-glutamine on Vital Signs - Respiration | Baseline to 48 weeks (12 months)
  Patient's respiration will be collected at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka L Niihara, MD, Study Chair — Emmaus Medical, Inc.
Locations (3):
- United States (3):
  - The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Ventura Clinical Trials, Ventura, California
  - Clinical Trials of Texas, Inc., San Antonio, Texas